CLINICAL TRIAL: NCT07106333
Title: Management of Post-Extraction Localized Alveolar Osteitis
Brief Title: Assessment of Ozone Therapy for Management of Post-Extraction Localized Alveolar Osteitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohammed El-Sawy, Clinical Professor and principle investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADMNF-00225
Record Dates: First submitted 2025-07-15; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Alveolar Osteitis
MeSH Terms: conditions — Dry Socket | interventions — Therapeutic Irrigation; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: intervention after wisdom tooth extraction either with saline or with topical ozone
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Conventional Treatment (Control Group): (Other): Socket debridement and irrigation with normal saline.
  Pain management using Diclofenac potassium (50 mg TID).
  Follow-up at day 2, 3, 7, 10, and 14.
  Home care: saline mouth rinse.
  Interventions: Other: Irrigation with saline
- Group B-Ozone Therapy Group (Other): Socket debridement and irrigation with ozonated water.
  Application of ozonated gel into the socket using syringe with fine-tip applicator.
  Pain management using Diclofenac potassium (50 mg TID).
  Patients instructed to use ozonated water and gel at home daily.
  Follow-up at day 2, 3, 7, 10, and 14.
  Interventions: Other: Topical Ozone Therapy

INTERVENTIONS:
Other: Topical Ozone Therapy — The intervention involves local application of ozone in two forms:
  Ozonated Water - used for irrigation of the extraction socket.
  Ozonated Gel - applied topically inside the socket to promote healing and reduce pain.
  Both are used after socket debridement and bleeding provocation, followed by standard analgesic administration (Diclofenac potassium).
  Arms: Group B-Ozone Therapy Group
Other: Irrigation with saline — The intervention involves irrigation with saline
  Arms: Group A - Conventional Treatment (Control Group):

SUMMARY:
This clinical study investigates the effectiveness of ozone therapy in comparison to conventional treatment for alveolar osteitis (AO), a common painful complication following tooth extraction. Forty patients diagnosed with dry socket will be randomly divided into two groups. Group A will receive traditional treatment with normal saline irrigation and analgesics, while Group B will be treated using ozonated water, ozonated gel, and analgesics. Both groups will be monitored over a two-week period to evaluate pain levels, healing progression, and other clinical indicators. The study aims to assess the palliative and regenerative benefits of ozone therapy in managing AO, potentially offering an alternative to conventional symptomatic treatments.

DETAILED DESCRIPTION:
Alveolar osteitis (AO), commonly referred to as "dry socket," is a frequent postoperative complication following tooth extraction. It typically presents 1-3 days post-extraction with severe pain due to premature loss or breakdown of the blood clot within the extraction socket. While the exact pathogenesis remains controversial, enhanced fibrinolytic activity, bone trauma, and bacterial contamination are considered primary contributing factors. The incidence is notably higher in mandibular third molars.

Traditional management approaches-such as saline irrigation, antibiotics, and eugenol-based dressings-are often palliative and do not directly target the underlying cause. Ozone therapy, with its antimicrobial, analgesic, and wound-healing properties, has recently emerged as a potential alternative. Ozone, when applied in water or gel forms, is believed to promote clot stability, reduce pain, and enhance soft tissue regeneration.

Aim of the Study:

To assess and compare the palliative (pain-relieving) and regenerative (healing-promoting) effects of ozone therapy versus conventional treatment in patients suffering from alveolar osteitis.

ELIGIBILITY:
Inclusion Criteria:

Age: 18-60 years.

Patients undergoing simple (non-surgical) extractions.

Medically healthy individuals.

Exclusion Criteria:

Patients already treated for AO.

Presence of systemic diseases affecting healing.

Severe infections or facial swelling.

Incomplete follow-up.

Contraindications to ozone therapy: G6PD deficiency, hyperthyroidism, malignant hypertension, recent myocardial infarction.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction | Pain intensity will be recorded at: Day 2 Day 3 Day 7 Day 10 Day 14
  Patient-reported pain scale, categorized as:
  Severe
  Moderate
  Mild
  No pain

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed El-Sawy, PhD, Study Chair — Menoufia Universityt

IPD SHARING:
Plan to Share IPD: No
Up on request from the corresponding author